CLINICAL TRIAL: NCT03687203
Title: Cognitive-driven ADL Impairment as a Predictor for Parkinson's Disease Dementia (PDD)
Brief Title: Cognitive-driven ADL Impairment as a Predictor for PDD
Status: Completed | Type: Observational
Sponsor: University Hospital Tuebingen (Other)
Collaborators: Sub-Investigator, Dr. Kathrin Brockmann, University Hospital of Tuebingen, Tuebingen, Germany (Unknown); Advisory board, Prof. Dr. Thomas Gasser, University Hospital of Tuebingen, Tuebingen, Germany (Unknown); Advisory board, Prof. Dr. Berg, Christian-Albrechts-University, Kiel, Germany (Unknown)
Responsible Party: Principal Investigator, PD Dr. Inga Liepelt-Scarfone, PhD, University Hospital Tuebingen
Other Study IDs: 284/2018BO1
Record Dates: First submitted 2018-09-20; First posted 2018-09-27 (Actual); Last update posted 2022-02-24 (Actual); Status verified 2021-01

CONDITIONS: Parkinson Disease
Keywords: Activity of daily living function; Cognitive impairment; Parkinson's disease dementia
MeSH Terms: conditions — Parkinson Disease; Cognitive Dysfunction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Through venipuncture, the following samples will be taken:
  * venous blood for the determination of routine values (1 Serum tube)
  * venous blood for RNA Isolation
  * venous blood for DNA isolation
  * venous blood in 1 Serum tube
  A lumbar puncture at level L3/L4 or L4/L5 of the spine will be performed by a qualified clinician in subsample of the cohort. Neurodegenerative markers such as Abeta1-42 and Abeta1-40 will be analysed.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Functional Activities Questionnaire — The FAQ is an economic and easy to apply activity of daily living scale. We aim to validate the prognostic value of novel FAQ scores, which differentiate cognitive- from motor-driven activity of daily living function.

SUMMARY:
Mild cognitive impairment in Parkinson's disease (PD-MCI) is the highest risk factor for Parkinson's disease dementia (PDD). The core feature for differentiating PDD from PD-MCI is the loss of the ability to perform activities of daily living (ADL). As Parkinson's Disease (PD) is primarily a movement disorder, the distinction between motor and cognitive contributions to ADL in PD is an obvious challenge, which the investigators aimed to explore in this study. The goal of the study is to evaluate whether PD-MCI patients with more pronounced, cognitive-driven ADL impairment are at higher risk for cognitive worsening and PDD. A longitudinal follow-up assessment of 262 non-demented PD patients will be conducted over the next two years, with a comprehensive clinical assessment as well as biomarker sampling (cerebrospinal fluid and blood markers). Primary longitudinal outcome will be conversion to PDD and PD-MCI. Conversion rates of patients with and without additional mild cognitive-driven ADL impairment at baseline will be compared. Novel scores of the Pfeffer Functional Activities Questionnaire (FAQ) are used to assess instrumental ADL, differentiating between cognitive- and motor-driven ADL impairment in PD-MCI.

ELIGIBILITY:
Inclusion Criteria:

* Participation in the baseline assessment
* Ability to communicate well with the investigator, to understand and comply with the requirements of the study.
* Provide written informed consent to participate in the study and understand their right to withdraw consent at any time without prejudice to future medical care.

Exclusion Criteria:

* Any disability that may prevent the subject from completing the informed consent form or other study requirements.
* Other neurodegenerative disease which renders the subject unable to communicate well with the investigator or to understand and comply with the requirements of the study.
* Participation in any clinical investigation of a new investigational compound or therapy within 4 weeks prior to baseline visit, and for any other limitation of participation based on local regulations.
* Alcohol, medication or drug dependency or abuse (except for nicotine).
* History of brain disease other than PD, e.g. head trauma, stroke, encephalitis, etc.

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants of the already recruited ABC-PD (Amyloid-Beta in cerebrospinal fluid as a risk factor for cognitive dysfunction in Parkinson's Disease) cross-sectional cohort (Ethic Protocol of the Medical Faculty Tuebingen 686/2013B01) will be asked to participate in the follow-up assessment. A drop-out rate of 20% is expected for follow-up retention. Therefore, investigation of 209 patients will be conducted between August 2018 and April 2020.
Sampling Method: Non-Probability Sample
Enrollment: 182 (Actual)
Dates: Start 2018-07-20 (Actual); Primary Completion 2020-10-15 (Actual); Study Completion 2021-01-31 (Actual)

PRIMARY OUTCOMES:
Functional Activity Questionnaire | 8 minutes
  Assessment of cognitive- and motor driven activity of daily living function

CONTACTS AND LOCATIONS:
Overall Officials: Inga Liepelt-Scarfone, PhD, Principal Investigator — University Hospital Tuebingen
Locations (1):
- University hospital of Tuebingen, Tübingen, Baden-Wurttemberg, Germany

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Becker S, Bode M, Brockmann K, Gasser T, Michaelis K, Solbrig S, Nuerk HC, Schulte C, Maetzler W, Zimmermann M, Berg D, Liepelt-Scarfone I. Cognitive-Driven Activities of Daily Living Impairment as a Predictor for Dementia in Parkinson Disease: A Longitudinal Cohort Study. Neurology. 2022 Dec 5;99(23):e2548-e2560. doi: 10.1212/WNL.0000000000201201. PMID 36240089

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-07-05): https://cdn.clinicaltrials.gov/large-docs/03/NCT03687203/Prot_SAP_000.pdf